CLINICAL TRIAL: NCT03356626
Title: Comparison of Perioperative Outcomes Between Bipolar Sealing Device and Ultrasonic Shears During Laparoscopic Gastrectomy for Early Gastric Cancer
Brief Title: Comparison of Perioperative Outcomes Between Energy Device During Laparoscopic Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Medtronic Spine LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: EBD-02
Record Dates: First submitted 2017-11-24; First posted 2017-11-29 (Actual); Results first posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2022-05

CONDITIONS: Postoperative Inflammation; Postoperative Fever
Keywords: fever, inflammation
MeSH Terms: conditions — Fever; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ULTRACISION Harmonic Scalpel (Experimental): Patients group randomized to use ULTRACISION Harmonic Scalpel when receives laparoscopic gastrectomy
  Interventions: Device: ULTRACISION Harmonic Scalpel
- Ligasure Maryland (Experimental): Patients group randomized to use Ligasure Maryland when receives laparoscopic gastrectomy
  Interventions: Device: Ligasure Maryland
- Thunderbeat (Experimental): Patients group randomized to use Thunderbeat when receives laparoscopic gastrectomy
  Interventions: Device: Thunderbeat

INTERVENTIONS:
Device: ULTRACISION Harmonic Scalpel — to use ULTRACISION Harmonic Scalpel when performing gastrectomy
  Arms: ULTRACISION Harmonic Scalpel
Device: Ligasure Maryland — to use Ligasure Maryland when performing gastrectomy
  Arms: Ligasure Maryland
Device: Thunderbeat — to use Thunderbeat when performing gastrectomy
  Arms: Thunderbeat

SUMMARY:
To find out which instrument can be much better for laparoscopic gastrectomy among Harmonic scalpel, Ligasure Maryland, Thunderbeat

comparing postoperative CRP level in each group

DETAILED DESCRIPTION:
To find out which instrument can be much better for laparoscopic gastrectomy among Harmonic scalpel, Ligasure Maryland, Thunderbeat

comparing postoperative CRP level in each group

1. post operative 2nd day CRP level
2. post operative 4th day CRP level
3. post operative IL-6, 10 level in 2nd, 4th day

ELIGIBILITY:
Inclusion Criteria:

* pathologically proven adenocarcinoma in stomach
* patients who are expected for R0 resection with distal gastrectomy
* pre-operative clinical stage should be stage I
* patients who is able to be followed up with in postoperative 30 days
* patients whose CRP is normal before surgery

Exclusion Criteria:

* patients who had an abdominal surgery
* patients who received chemotherapy, radiotherapy before surgery
* patients who received ESD before surgery
* Patients who had an ascites on pre-operative CT scan
* liver cirrhosis
* cardiovascular disease (Ejection Fraction<50%)
* serum creatinine > 1.4 mg/dL or BUN>26mg/dL
* PT INR >1.2 or aPTT>45sec
* uncontrolled diabetes
* Crohn's disease, ulcerative colitis
* patients who receives anti-coagulants
* patients who need pre-operative steroid booster because of steroid treatment
* pregnancy
* patients who have allergic reaction to iodine

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2021-01-07 (Actual); Study Completion 2022-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seong-Ho Kong, MD,PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Groups:
- ULTRACISION Harmonic Scalpel: Patients group randomized to use ULTRACISION Harmonic Scalpel when receives laparoscopic gastrectomy ULTRACISION Harmonic Scalpel: to use ULTRACISION Harmonic Scalpel when performing gastrectomy
- Ligasure Maryland: Patients group randomized to use Ligasure Maryland when receives laparoscopic gastrectomy Ligasure Maryland: to use Ligasure Maryland when performing gastrectomy
- Thunderbeat: Patients group randomized to use Thunderbeat when receives laparoscopic gastrectomy Thunderbeat: to use Thunderbeat when performing gastrectomy
Period: Overall Study
Arm/Group | ULTRACISION Harmonic Scalpel | Ligasure Maryland | Thunderbeat
Started | 61 | 65 | 63
Completed | 57 | 60 | 57
Not Completed | 4 | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ULTRACISION Harmonic Scalpel | Ligasure Maryland | Thunderbeat | Total
Number analyzed (Participants) | 57 | 60 | 57 | 174
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.75 (11.01) | 60.35 (11.01) | 62.51 (10.00) | 61 (10.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 26 | 14 | 52
  Male | 45 | 34 | 43 | 122
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 57 | 60 | 57 | 174
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 57 | 60 | 57 | 174
Preoperative CRP level [Mean (Standard Deviation); unit: mg/dL] | 0.21 (0.18) | 0.16 (0.16) | 0.16 (0.14) | 0.18 (0.16)

OUTCOME MEASURES:

1. Primary Outcome: Postoperative 2nd Day CRP
Description: To check the postoperative 2nd day CRP level in each group
Time Frame: 2nd day
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | ULTRACISION Harmonic Scalpel | Ligasure Maryland | Thunderbeat
Number analyzed (Participants) | 57 | 60 | 57
mg/dL | 11.12 (5.02) | 9.03 (5.55) | 12.67 (6.14)

2. Secondary Outcome: Postoperative 4th Day CRP
Description: To check the postoperative 4th day CRP level in each group
Time Frame: 4th day
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | ULTRACISION Harmonic Scalpel | Ligasure Maryland | Thunderbeat
Number analyzed (Participants) | 57 | 60 | 57
mg/dL | 9.62 (0.53) | 7.48 (0.52) | 9.48 (0.53)

3. Secondary Outcome: Postoperative 2nd Day IL-6
Description: To check the postoperative 2nd, 4th day IL-6, IL10 level in each group
Time Frame: 2nd day
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | ULTRACISION Harmonic Scalpel | Ligasure Maryland | Thunderbeat
Number analyzed (Participants) | 57 | 60 | 57
pg/ml | 17.96 (3.82) | 19.32 (3.51) | 22.3 (3.61)

4. Secondary Outcome: Postoperative 4th Day IL-6
Description: To check the postoperative 2nd, 4th day IL-6, IL10 level in each group
Time Frame: 4th day
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | ULTRACISION Harmonic Scalpel | Ligasure Maryland | Thunderbeat
Number analyzed (Participants) | 57 | 60 | 57
pg/ml | 8.08 (3.82) | 8.07 (3.62) | 7.16 (3.61)

5. Secondary Outcome: Postoperative 2nd Day IL-10 Level
Description: To check the postoperative 2nd, 4th day IL-6, IL10 level in each group
Time Frame: 2nd day
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | ULTRACISION Harmonic Scalpel | Ligasure Maryland | Thunderbeat
Number analyzed (Participants) | 57 | 60 | 57
pg/ml | 3.52 (0.04) | 3.53 (0.04) | 3.49 (0.04)

6. Secondary Outcome: Postoperative 4th Day IL-10 Level
Description: To check the postoperative 2nd, 4th day IL-6, IL10 level in each group
Time Frame: 4th day
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | ULTRACISION Harmonic Scalpel | Ligasure Maryland | Thunderbeat
Number analyzed (Participants) | 57 | 60 | 57
pg/ml | 0.47 (0.71) | 0.47 (0.71) | 0.52 (0.66)

ADVERSE EVENTS:
Time Frame: 30 days after operation
Arm/Group | ULTRACISION Harmonic Scalpel | Ligasure Maryland | Thunderbeat
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/60 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/60 | 0/57
Other Adverse Events (participants affected / at risk) | 2/57 | 3/60 | 4/57
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ULTRACISION Harmonic Scalpel (N=57) | Ligasure Maryland (N=60) | Thunderbeat (N=57)
Postoperative complication: Clavien-Dindo grade < IIIa (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Postoperative complication: Clavien-Dindo grade ≥ IIIa † (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3)

LIMITATIONS AND CAVEATS:
The complication rate, could not be evaluated due to the limited number of cases. A stratified randomization method was chosen in this study to prevent an imbalance of prognostic factors that could affect the results, but the baseline characteristics of the patients in each group were not perfectly balanced. Since gastric surgery may be affected by patient factors, such as sex and BMI, those factors should be considered stratification factors.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/26/NCT03356626/Prot_SAP_000.pdf